CLINICAL TRIAL: NCT06576934
Title: Early Implantation of a Transjugular Intrahepatic Portosystemic Shunt (TIPS) in Patients With Liver Cirrhosis and Ascites: a Multicentre, Randomised Controlled Trial
Brief Title: Early TIPS in Patients With Liver Cirrhosis and Ascites
Acronym: eTIPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Jena University Hospital (Other); Johannes Gutenberg University Mainz (Other); University Hospital Muenster (Other); University Hospital, Bonn (Other); University Hospital Munich (LMU) (Unknown); Hannover Medical School (Other); University of Leipzig (Other); University Hospital, Aachen (Other); University Hospital Lübeck (Other); Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dominik Bettinger, Principal Investigator, University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: eTIPS
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Liver Cirrhosis; Ascites Hepatic; Portal Hypertension
Keywords: liver cirrhosis; Transjugular intrahepatic portosystemic shunt; ascites; MELD
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Ascites | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transjugular intrahepatic portosystemic shunt (TIPS) (Experimental): Patients will receive TIPS implantation if ascites as the first single decompensating event with grade 2 ascites and MELD ≥ 15 OR grade 3 ascites occurs.
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunt (TIPS)
- Standard medical treatment (No Intervention): Patients in this group will receive standard medical treatment according to the current EASL guidelines (salt restriction, diuretic treatment, carvedilol, large-volume paracentesis if necessary, albumin substitution if more than 5 litre of ascites is removed)

INTERVENTIONS:
Procedure: Transjugular intrahepatic portosystemic shunt (TIPS) — TIPS implantation is performed by creating a shunt between the liver vein and the portal vein to enable portal pressure reduction.
  Arms: Transjugular intrahepatic portosystemic shunt (TIPS)

SUMMARY:
The aim of this clinical trial is to compare the safety and efficacy of transjugular intrahepatic portosystemic shunt (TIPS) implantation with standard treatment (diuretic medications, and if necessary, paracenteses) in patients with liver cirrhosis and development of ascites as the first decompensating event.

By creating a shunt between the liver vein and the portal vein, blood is diverted from the portal vein directly into the hepatic vein, which results in a reduction of pressure in the portal vein so that development of ascites is reduced.

DETAILED DESCRIPTION:
Complications in patients with liver cirrhosis are mainly due to the development of clinical significant portal hypertension. These complications include development of varices and ascites. Implantation of a transjugular intrahepatic portosystemic shunt (TIPS) has emerged as a safe and effective interventional treatment of portal hypertension. TIPS implantation is recommended for secondary prophylaxis of variceal bleeding. Further, in patients with acute variceal bleeding, early TIPS implantation within 72 hours after the bleeding episode is associated with a lower re-bleeding rate and also improved survival in high risk patients. In patients with ascites, TIPS implantation is recommend in more advanced stages when conservative treatment has failed to control ascites. Importantly, ascites clearance can be achieved in only 51% in these patients. Recently, it has been shown that patients with a lower paracenteses frequency have a higher chance of ascites control compared to patients with long-term paracenteses. These data suggest that TIPS implantation in patients with ascites should not be delayed comparable to patients with acute variceal bleeding. The presented study aims to analyse the concept of early TIPS implantation in patients with liver cirrhosis and ascites.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this trial must meet all of the following criteria:

1. Patients ≥ 18 years and < 80 years
2. Liver cirrhosis as documented by previous liver biopsy or by a combination of typical clinical, biochemical and sonographic features
3. Ascites as the first single decompensating event with grade 2 ascites and MELD ≥ 15 OR grade 3 ascites
4. INR ≤ 1.5
5. Ability to understand the nature of the trial and the trial related procedures and to comply with them

Exclusion Criteria:

Patients eligible for this trial must not meet any of the following criteria:

1. Treatment refractory or recurrent ascites at the time of study inclusion
2. Patients with concomitant variceal bleeding fulfilling the criteria for pre-emptive TIPS implantation (Child-Pugh class C < 14 points or Child-Pugh class B >7 with active bleeding at initial endoscopy or hepatic venous pressure gradient [HVPG] > 20 mmHg at the time of bleeding)
3. Budd-Chiari syndrome
4. Portal vein thrombosis (PVT)
5. Spontaneous bacterial peritonitis (SBP)
6. Uncontrolled systemic infection (defined as an increase of > 20% if inflammatory parameters [C-reactive protein, procalcitonin, leukocytes] and/or sepsis as a reason for development of ascites
7. Cardiac cirrhosis (defined as the development of liver cirrhosis in a patient with cardiac heart failure due to primary cardiac disease)
8. Clinical significant cardiac disease (NYHA ≥II)
9. Untreated valvular heart disease: middle to high-grade valve stenosis or insufficiency (applies to mitral, tricuspid, aortic and pulmonary valves)
10. Diastolic dysfunction grade III, stated by transthoracic echocardiogram (TTE)
11. Reduced left ventricular ejection fraction ≤50%
12. Pulmonary hypertension (mean pulmonary arterial pressure > 45 mmHg)
13. Bilirubin > 3 mg/dl
14. Obstructive cholestasis
15. Hepatorenal syndrome type AKI (HRS-AKI)
16. Acute on chronic liver failure
17. Benign liver tumor within the potential puncture tract
18. Patient after liver transplantation
19. Prior TIPS implantation
20. Ongoing and/or recurrent hepatic encephalopathy (grade >II)
21. Active tumor disease including hepatocellular carcinoma defined as need for chemotherapy, radiation therapy, interventional or surgical treatment
22. New onset of antiviral treatment for chronic hepatitis B virus (HBV) infection within the last 3 months
23. Untreated chronic hepatitis C virus (HCV) infection
24. Life expectancy <1 year
25. Pregnant or breastfeeding women
26. Patients without the legal capacity who are unable to understand the nature, significance and consequences of the study
27. Simultaneous participation in other interventional trials which could interfere with this trial; simultaneous participation in registry and diagnostic trials is allowed
28. Person who is in a relationship of dependence/employment with the sponsor or the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Transplantation-free survival (TFS) | Through study completion, an average of 12 months
  The primary objective of this study is to assess a survival benefit in patients with early allocation to TIPS implantation in comparison to patients with standard medical treatment (SMT).

SECONDARY OUTCOMES:
Time to ascites with need for paracenteses | Through study completion, an average of 12 months
  Assessment of the duration until the next paracentesis after randomisation occurs to compare the efficacy of TIPS implantation compared to standard medical treatment.
Assessment of quality of life | Through study completion, an average of 1 year: at study inclusion, at 6 and 12 months after randomisation
  Quality of life assessed with the SF-36 and CLDQ (chronic liver disease questionnaire) before TIPS implantation/study inclusion, 6 and 12 months after randomisation.
Rate of TIPS implantation in the standard medical treatment group | Through study completion, an average of 12 months
  Need for TIPS implantation (recurrent ascites or variceal bleeding) in the standard medical treatment group.
Rate of TIPS dysfunction | Through study completion, an average of 12 months
  Development of TIPS dysfunction in the TIPS group

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bettinger D, Janoschke M, Jenkner C, Kaufmann M, van Gessel J, Otter HH, Schultheiss M, Thimme R; on behalf of the eTIPS study group. Early implantation of a transjugular intrahepatic portosystemic shunt (TIPS) in patients with liver cirrhosis and ascites (eTIPS): a multicentre, randomised controlled trial. Trials. 2025 Oct 2;26(1):385. doi: 10.1186/s13063-025-09038-8. PMID 41039580